CLINICAL TRIAL: NCT02986646
Title: Comparison of Intra-articular and Intra-tendinous Injections for Treatment of Lateral Epicondylitis: A Randomized, Controlled Trial
Brief Title: Comparison of Intra-articular and Intra-tendinous Injections for Treatment of Lateral Epicondylitis
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Akin Cil, Franklin D. Dickson Associate Professor, Vice Chairman, Department of Orthopaedic Surgery, Truman Medical Centers, University of Missouri, Kansas City
Other Study IDs: 16-280; 17-022 (Other: Truman Medical Center)
Record Dates: First submitted 2016-11-17; First posted 2016-12-08 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- physical therapy (PT) and rest: This group of subjects will be prescribed a physical therapy home exercise program and rest (of the injured elbow).
- PT and intra-tendinous steroid injection: This group of subjects will be prescribed a physical therapy home exercise program and will received an intra-tendinous corticosteroid injection into the area of the ECRB origin (of the injured elbow).
- PT and intra-articular steroid injection: This group of subjects will be prescribed a physical therapy home exercise program and will received an intra-articular corticosteroid injection into the elbow joint (of the injured elbow).

SUMMARY:
Lateral epicondylitis, commonly known as "tennis elbow" is a common cause of elbow pain encountered in primary care and specialty clinics. Although lateral epicondylitis is common, little consensus exists on the best way to treat it. Historically 80% of patients will get better with non-operative treatments (rest, NSAIDS, bracing and injections). In regard to efficacy of injections, recent large, prospective, randomized studies have shown minor improvements in the short term, but no long term benefits when compared to saline injection. Consistently, intra-articular injections have not been reported. The investigators suspect that elbow joint inflammation may be an underappreciated source of pain in lateral epicondylitis. The investigators' hypothesis is that patients receiving intra-articular injections will have greater improvement compared to patients receiving either no injection or an intra-tendinous injection.

DETAILED DESCRIPTION:
Background Lateral epicondylitis, commonly known as "tennis elbow" is a common cause of elbow pain, occurring in 1-3% of adults each year. It is a common pathology encountered in primary care, as well as specialty clinics. The typical patient is in his or her 4th-5th decade. Males and females are affected equally and the dominant arm is more commonly involved. Patients participating in sports or work related activities involving repetitive forearm rotation with the elbow extended are at high risk for developing symptoms. Symptom onset is insidious and related to repetitive microtrauma, similar to other chronic overuse tendinopathies. Patients classically present with tenderness over the lateral aspect of the elbow, just distal and anterior o the lateral epicondyle, at the origins of the extensor carpi radialis brevis (ECRB) and the extensor digitorum communis (EDC) muscles. Pain is worsened with resisted wrist and finger extension. 1,2 Much of the information the investigators have regarding the lateral epicondylitis is from the work of Nirschl and colleagues. The etiology of lateral epicondylitis is believed to result from small tears of the ECRB origin from repetitive microtrauma. Gross examination reveals grayish, immature scar tissue that appears shiny, edematous and friable. Histologic analysis reveals what has been termed "angiofibroblastic hyperplasia" of the ECRB tendon origin. There are no inflammatory cells noted on histology, putting into question the classification of lateral epicondylitis as an inflammatory condition.3-6 Baker et al have noted consistent capsular changes seen on arthroscopy and developed a classification system, hinting that another source of pain may be inside the joint.7,8 Early authors described a mass of grayish tissue under the ECRB origin, intimate with the joint capsule. It may be that this tissue causes capsular inflammation, leading to elbow pain.9 Although lateral epicondylitis is common, little consensus exists on the best way to treat it. Historic teaching is that 80% of patients will get better with non-operative treatments, ranging from relative rest, NSAIDs, bracing and injections. There will be approximately 4-11% of patients, however, that will require operative treatment before symptom resolution.1 Current mainstays of treatment are non-operative. Many patients do get better with rest and activity avoidance. Counterforce braces do not lead to quicker recovery, however, they do allow for more forceful activity during that recovery period.10 NSAIDs have not shown added benefit long term either.1,2 There has been significant interest in the efficacy of injections in treatment of both acute and chronic lateral epicondylitis. Steroid injections have been used as standard treatment for decades. Anecdotally, patients do well with injections. Recent large, prospective, randomized studies have shown minor improvements in the short term, but no long term benefits when compared to saline injection.11-15 Protocols for these studies varied greatly, both in steroid utilized and injection technique. Common injection techniques included injecting at the point of maximal tenderness versus at the ECRB origin. Additionally, some authors injected a single time, whereas others used a peppering technique, with one skin entry point and multiple entry points in the muscle. Consistently, however, no intra-articular injections were reported. The investigator suspect that elbow joint inflammation may be an underappreciated source of pain in lateral epicondylitis. Our hypothesis is that patients receiving intra-articular injections will have greater improvement compared to patients receiving either no injection or an intra-tendinous injection.

Statement of Objectives

1. To directly compare outcomes of patients with lateral epicondylitis who receive one of three treatment options: 1. physical therapy and rest 2. physical therapy and intra-tendinous corticosteroid injection or 3. physical therapy and intra-articular corticosteroid injection.
2. To blind both patient and assessing physician/nurse research coordinator to the treatment that was received for the duration of the study, in order to reduce the effect of any potential bias.
3. To collect outcome data, both subjectively from the patient using proven outcome measures, and objectively from regularly spaced follow up visits with blinded assessors.
4. To collect and comment on data from the three treatment groups regarding outcomes related to pain scores, functional outcomes and recurrence of symptoms.

Materials & Methods This will be a randomized, double-blind, controlled trial comparing patients who receive physical therapy and rest, physical therapy and intra-tendinous corticosteroid injection or physical therapy and intra-articular corticosteroid injection for the treatment of lateral epicondylitis. To our knowledge there are no level I or II studies evaluating intra-articular elbow injections in the literature. All patients will be treated at one hospital system at one of 2 locations Truman Medical Center-Hospital Hill (TMC-HH) or Truman Medical Center- Lakewood (TMC-LW), by the principal investigator Our goal is to enroll patients who are seeking care from either a primary care sports medicine physician or orthopaedic surgeon for their persistent and limiting elbow pain. Potential subjects who meet inclusion criteria will be approached about participating in the study. Enrollment will continue until sufficient numbers have been reached to determine a significant difference. Based on our power analysis a total of 82 patients will be enrolled in the study.

Lateral epicondylitis is a clinical diagnosis.1,2 In our patients, diagnosis will be made based on a thorough history and physical examination. Patients with lateral epicondylitis are typically present in the 4th or 5th decade of life with vague, lateral elbow pain. The pain is of insidious onset without a singular inciting event. Symptoms are typically in the dominant arm and occur in patients that perform activities involving repeated wrist extension against resistance. Patients typically do not have mechanical symptoms as is seen with loose bodies or osteochondral lesions. Neurologic deficits or alterations are not seen with this condition. Systemic inflammatory diagnoses, such as rheumatoid arthritis or systemic lupus erythematosus can have widespread vague joint pains that can confound the diagnosis of lateral elbow pain. Patients with these conditions will be excluded.

On physical examination, patients will have tenderness about the lateral elbow, typically at the origin of the ECRB tendon just distal to the lateral epicondyle. This pain will be exacerbated by resisted extension of the wrist, and/or resisted extension of the long finger. In rare cases elbow ROM will be limited. Standard elbow radiographs will be obtained to rule out fracture, arthritis, intra-articular loose body, deformity, osteonecrosis, osteochondral lesion, neoplasm and subtle instability. Posterolateral rotatory instability (PLRI) of the elbow is another source of lateral elbow pain, and posterolateral drawer testing will be performed on all patients to rule out this condition. Although cubital tunnel syndrome typically causes medial elbow pain, it can present with non-focal, vague pain. A combination of a thorough neurologic exam of the distal extremity along with compression of the cubital tunnel and presence or absence of a Tinel's sign at the elbow will be used to diagnosis the presence of this condition. Patients who have concern for shoulder or wrist pathology or cervical spine pathology will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of lateral epicondylitis based on 2 or more of the following diagnostic criteria: tenderness over the lateral epicondyle; pain with resisted wrist extension; pain with resisted long finger extension.
* Symptoms lasting a minimum of 6 weeks
* Pain score of >= 3/10 using the Visual Analog Scale (VAS)
* Age >= 18 years

Exclusion Criteria:

* History of prior elbow surgery
* History elbow fracture within the past year
* Elbow instability on physical examination
* Elbow arthritis on radiographs
* Compressive neuropathy in the affected extremity (i.e.carpal tunnel, cubital tunnel)
* Evidence of cervical myelopathy, radiculopathy or brachial plexopathy
* History of systemic inflammatory condition (i.e. rheumatoid arthritis or systemic lupus erythematosus)
* Allergy to study administered medications (steroid or lidocaine)
* Neoplasm
* Non-English speaking patients
* Inability to comply with study protocols and follow up.
* Pregnant female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are seeking care from either a primary care sports medicine physician or orthopaedic surgeon for their persistent and limiting elbow pain.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-01; Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
PRTEE (Patient Rated Tennis Elbow Evaluation) | 2 years
  The primary analysis will compare the PRTEE scores of each group at 2 years post-enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Akin Cil, Principal Investigator — University of Missouri Kansas City, Department of Orthopaedic Surgery
Locations (1):
- Truman Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No